CLINICAL TRIAL: NCT01693497
Title: Comparison of a Gestalt-based Approach to PTSD Therapy With Cognitive Processing Therapy
Brief Title: Comparison of Cognitive Processing Therapy (CPT) and Dialogical Exposure Therapy (DET) for Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Willi Butollo, Head of Clinical Psychology and Psychotherapy, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gestalt therapy for PTSD
Record Dates: First submitted 2012-09-18; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; PTSD; psychotherapy; randomized trial; gestalt
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dialogical exposure therapy (Experimental): Psychotherapy based on a manual integrating Gestalt principles with cognitive-behavioral techniques.
  Interventions: Behavioral: Dialogical exposure therapy
- Cognitive Processing Therapy (Active Comparator): Cognitive Processing Therapy, a cognitive behavioral psychotherapy for PTSD patients. Based on a German manual adapted from Resick and Schnicke, 1993.
  Interventions: Behavioral: Cognitive Processing Therapy (German Adaptation)

INTERVENTIONS:
Behavioral: Dialogical exposure therapy — This 24-session treatment protocol includes cognitive-behavioral components integrated with a frame based on gestalt principles. There are four phases, safety, stabilization, confrontation and integration.
  Arms: Dialogical exposure therapy
Behavioral: Cognitive Processing Therapy (German Adaptation) — This is a German adaptation of Cognitive Processing Therapy, developed by Prof. P. A. Resick. This intervention includes cognitive restructuring, a focus on the traumatic memory and a focus on issues that are likely to be problematic in traumatized individuals.
  Arms: Cognitive Processing Therapy

SUMMARY:
This study aims to compare two active psychological treatments for PTSD. One is an established therapy, Cognitive Processing Therapy (CPT) which operates as a control condition for a newly developed intervention, an integrative Gestalt-based trauma therapy, Dialogical Exposure Therapy (DET). There is no inactive control condition. We expect the two therapies to perform on a similar level, which would constitute evidence for the efficacy of DET.

ELIGIBILITY:
Inclusion Criteria:

* main diagnosis of posttraumatic stress disorder
* time since trauma is at least three months

Exclusion Criteria:

* acute suicidal ideation
* severe personality pathology
* substance dependence
* early childhood trauma (e.g. child sexual abuse)
* history of psychosis
* dissociative identity disorder
* neurological impairment (e.g. craniocerebral injury with functional impairment)
* severe pre-traumatic depression
* ongoing psychotherapy
* lack of motivation
* lack of German language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2002-09; Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
PTBS Symptom Severity | change from pretreatment to posttreatment (planned duration 12 weeks on average) to follow-up (six months after posttreatment)
  Even though participants are assessed by a clinical interview before entering the study, the primary outcome measure is the PDS which is applied before and after treatment as well as at 6-month follow-up.

SECONDARY OUTCOMES:
PTSD Symptom change (IES-R) | change from pretreatment to posttreatment (planned duration 12 weeks on average) to follow-up (six months after posttreatment). Also measured at each session (up to 24 time points between pre- and posttreatment).
  The IES-R is a short instrument for the measurement of PTSD symptom severity. In this study, the IES-R is applied before every session in order to measure symptom change over the time of the therapy.

OTHER OUTCOMES:
Brief Symptom Inventory | change from pretreatment to posttreatment (planned duration 12 weeks on average) to follow-up (six months after posttreatment)
  The Brief Symptom Inventory (BSI) is a measure of general psychological distress.
Inventory of Interpersonal Problems (IIP) | change from pretreatment to posttreatment (planned duration 12 weeks on average) to follow-up (six months after posttreatment)
  The IIP is a widely used instrument to measure interpersonal distress.

CONTACTS AND LOCATIONS:
Overall Officials: Willi Butollo, Prof., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- LS für Klinische Psychologie und Psychotherapie, Munich, Germany